CLINICAL TRIAL: NCT00281723
Title: Phase 2 Study of Efficacy of Adhesive Tablets in Treating Oral Ulcers (Aphthous)
Brief Title: Efficacy of Adhesive Tablets in Treating Oral Ulcers (Aphthous)
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: The company which holds the patent was not interested.
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Grant from "Axiomedic. Advanced Medical Solutions", Zurich, Switzerland (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6-12.2.06-HMO-CTIL
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2007-05-08 (Estimated); Status verified 2007-05

CONDITIONS: Ulcer, Aphthous
Keywords: Aphthous; oral
MeSH Terms: conditions — Stomatitis, Aphthous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Pro-Pe adhesive tablet

SUMMARY:
Recurrent Aphthous Stomatitis (RAS) of the oral mucosa is a common and painful condition. Despite advances in therapeutic means there is still necessary to find a way to alleviate the local pain and discomfort induced by the mucosal ulceration.

The hypothesis was to study the effectiveness and acceptance of a herbal adhesive tablets in the treatment of RAS.

Participants in the study will be examined for oral lesions, will be instructed how to apply the oral-tablet, and will be interviewed during the follow-up period up to one week after the application.

ELIGIBILITY:
Inclusion Criteria (in healthy individuals):

* Age above 18 years old.
* Non-pregnant women.
* Healthy or controlled chronic diseases.
* Examination at the Oral Medicine Clinic

Inclusion Criteria (in RAS patients):

* Age above 18 years old.
* Non-pregnant women.
* Clinical diagnosis of RAS.
* Examination at the Oral Medicine Clinic

Exclusion Criteria:

* Oral lesion suspected to be malignant.
* Ulcerative oral lesion other than RAS.
* Another experimental oral intervention within the last 24 hours.
* Pregnant women.
* Allergy to components of the Pro-pe adhesive tablet

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Study Completion 2007-05 (Estimated)

PRIMARY OUTCOMES:
Serial questionnaires within 1 week post treatment to assess patient's perception, patient's pain relief and local adverse events in comparison to his past experience with other local treatments for oral ulcers.

CONTACTS AND LOCATIONS:
Overall Officials: Rakefet Czerninski, DMD, Principal Investigator — Hebrew University-Hadassah School of Dental Medicine; Sharon Elad, DMD MSc, Principal Investigator — Hebrew University-Hadassah School of Dental Medicine
Locations (1):
- Hadassah Medical Organization,, Jerusalem, Israel

REFERENCES:
- [Background] Mizrahi B, Golenser J, Wolnerman JS, Domb AJ. Adhesive tablet effective for treating canker sores in humans. J Pharm Sci. 2004 Dec;93(12):2927-35. doi: 10.1002/jps.20193. PMID 15459950
- See also: Company website — http://www.axiomedic.com